CLINICAL TRIAL: NCT04908449
Title: A Comparison of the Analgesic Effects of Pectointercostal Fascial Plane Block (PIFB) Alone Versus PIFB With Rectus Sheath Block (RSB) in Cardiac Surgery: a Prospective, Randomized Controlled Trial.
Brief Title: Pectointercostal Fascial Plane Block (PIFB) Alone Versus PIFB With Rectus Sheath Block (RSB) in Cardiac Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Anne Castro, MD, Assistant Professor of Anesthesiology, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRO00040365
Record Dates: First submitted 2021-05-24; First posted 2021-06-01 (Actual); Results first posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Coronary Artery Disease; Postoperative Pain; Respiratory Failure
Keywords: local anesthetic; regional anesthesia; quality of recovery; postoperative pain; coronary artery bypass graft
MeSH Terms: conditions — Coronary Artery Disease; Pain, Postoperative; Respiratory Insufficiency | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Rectus sheath block block with PIFB (experimental arm) (Experimental): PIFB with local anesthetic with RSB with local anesthetic (bupivacaine)
  Interventions: Drug: Rectus sheath block with bupivacaine
- Rectus sheath block with PIFB (placebo arm) (Placebo Comparator): PIFB with local anesthetic with RSB placebo (saline)
  Interventions: Drug: Rectus sheath block with bupivacaine

INTERVENTIONS:
Drug: Rectus sheath block with bupivacaine — Rectus sheath block with local anesthetic versus sham block with saline
  Other Names: Rectus sheath block with saline placebo

SUMMARY:
The purpose of this study is to determine if ultrasound-guided bilateral pectointercostal fascial plane blocks with bilateral rectus sheath blocks block decrease pain scores, decrease opioid consumption, improve respiratory function, and improve quality of recovery in patients recovering from elective cardiac surgery involving primary median sternotomy and mediastinal chest tubes in comparison to pectointercostal fascial plane blocks alone.

DETAILED DESCRIPTION:
This is a single center, prospective, randomized, controlled, double-blinded study. We anticipate recruitment of 62 subjects, with 25-30 in each group.

Primary Outcomes:

Pain scores on a 0-10 visual analog scale (VAS) at rest and with deep breathing at 1, 3, 6, 12, 18, and 24 hours post-extubation between subjects receiving PIFB + RSB versus subjects receiving only PIFB.

Total cumulative opioid consumption at 24 and 48 hours post-operatively.

Secondary Outcomes:

* Intraoperative total opioid consumption
* Change from baseline on incentive spirometry at 1, 3, 12, and 24 hours post-extubation
* Time from ICU arrival to liberation from mechanical ventilation
* QoR-15 (Quality of Recovery) score23 24 hours after extubation
* Hospital and ICU length of stay

Preoperative Management :

Subjects will be randomized on the morning of surgery to receive bilateral PIFB and bilateral RSB with local anesthetic versus bilateral PIFB with local anesthetic and bilateral RSB with saline (placebo).

Intraoperative Management All subjects will receive the standard of care anesthetic regimen for their cardiac surgery.

Postoperative Management Each PIFB will be performed with 15 mL of 0.25% bupivacaine with 5 mcg/ml of epinephrine, and bilateral RSB will be performed with an additional 20 mL of 0.25% bupivacaine with 5 mcg/ml of epinephrine (10mL on each side).

Postoperative Evaluation:

Evaluation of acute postoperative pain intensity using a 0-10 visual analog scale (VAS) will be undertaken at the following time points, both at rest and with deep breathing:

• 1, 3, 6, 12, 18, and 24 hours post-extubation Incentive spirometry will be assessed at 1, 3, 12, and 24 hours post-extubation, with three measures taken at each time point in order to compare postoperative performance with baseline spirometry.

Review of the medical chart will be made post-operatively to gather other data, including total intraoperative oral morphine equivalent consumption, cumulative opioid consumption at 24 and 48 hours, time from ICU arrival to tracheal extubation, hospital and ICU length of stay, and QoR-15 (Quality of Recovery) score administered 24 hours after extubation (with margin of error of 18-30 hours to avoid waking patients in the middle of the night) . Occurrences of any adverse events reported by the subject or medical team will also be collected.

ELIGIBILITY:
Inclusion Criteria:

* Subjects scheduled for cardiac surgery involving primary median sternotomy and mediastinal chest tubes.
* Age 18-85 years of age
* BMI 18-50 kg/m2
* Weight > 60 kg

Exclusion Criteria:

* Left ventricular ejection fraction (LVEF) < 30%
* Preoperative, intraoperative, or immediate post-operative placement of intra-aortic balloon pump or deployment of extra-corporeal membrane oxygenation (ECMO)
* Inability to understand or speak English
* Allergy to bupivacaine or other amide local anesthetic
* Contraindication to peripheral nerve block (e.g. local infection, previous trauma to the block site)
* Chronic opioid consumption (daily oral morphine equivalent of >20 mg) in the past three months
* Severe pulmonary or hepatic disease
* Neurological deficit or disorder
* Suspected or known addiction to or abuse of illicit drug(s), prescription medicine(s), or alcohol within the past two years
* Uncontrolled anxiety, schizophrenia, or other severe psychiatric disorder

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2023-06-19 (Actual); Primary Completion 2024-11-08 (Actual); Study Completion 2024-11-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne Castro, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Rectus Sheath Block With PIFB (Experimental Arm): PIFB with local anesthetic with RSB with local anesthetic (bupivacaine)
  Rectus sheath block with bupivacaine: Rectus sheath block with local anesthetic versus sham block with saline
Period: Overall Study
Arm/Group | Rectus Sheath Block With PIFB (Experimental Arm) | Rectus Sheath Block With PIFB (Placebo Arm)
Started | 30 | 32
Completed | 30 | 30
Not Completed | 0 | 2
Not completed — Patient with major surgical bleeding unerlated to block | 0 | 1
Not completed — Patient required postop RVAD, unrelated to block | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Rectus Sheath Block With Pectointercostal Fascial Plane Block (Experimental Arm): PIFB with local anesthetic with RSB with local anesthetic (bupivacaine)
  Rectus sheath block with bupivacaine: Rectus sheath block with local anesthetic versus sham block with saline
- Rectus Sheath Block With Pectointercostal Fascial Plane Block (Placebo Arm): PIFB with local anesthetic with RSB placebo (saline)
  Rectus sheath block with bupivacaine: Rectus sheath block with local anesthetic versus sham block with saline
- Total: Total of all reporting groups
Arm/Group | Rectus Sheath Block With Pectointercostal Fascial Plane Block (Experimental Arm) | Rectus Sheath Block With Pectointercostal Fascial Plane Block (Placebo Arm) | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.5 (9.51) | 67.3 (8.79) | 67.42 (9.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 17
  Male | 22 | 21 | 43
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 30 | 30 | 60
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 60
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 28.9 (4.31) | 30.8 (6.17) | 29.82 (5.36)
Hypertension diagnosis [Count of Participants; unit: Participants] | 20 | 21 | 41
Diabetes diagnosis [Count of Participants; unit: Participants] | 8 | 7 | 15
Coronary artery disease diagnosis [Count of Participants; unit: Participants] | 23 | 25 | 48
Peripheral Vascular Disease diagnosis [Count of Participants; unit: Participants] | 3 | 3 | 6
Neuropathy diagnosis [Count of Participants; unit: Participants] | 2 | 4 | 6
Anxiety diagnosis [Count of Participants; unit: Participants] | 2 | 5 | 7
Depression diagnosis [Count of Participants; unit: Participants] | 4 | 5 | 9
History of Cerebral Vascular Accident [Count of Participants; unit: Participants] | 3 | 1 | 4
Chronic Kidney Disease/End Stage Renal Disease diagnosis [Count of Participants; unit: Participants] | 5 | 4 | 9
Chronic Obstructive Pulmonary Disease diagnosis [Count of Participants; unit: Participants] | 0 | 1 | 1
Coronary Artery Bypass Graft Surgery [Count of Participants; unit: Participants] | 18 | 20 | 38
Coronary Artery Bypass Graft with single valve [Count of Participants; unit: Participants] | 3 | 3 | 6
Single valve case [Count of Participants; unit: Participants] | 9 | 7 | 16
Aortic crossclamp time (hours) [Mean (Standard Deviation); unit: hours] — The block occurred at the end of surgery, so in no way should have affected intraoperative surgical characteristics. The characteristics of surgery are therefore a baseline measure, not an outcome measure.
  hours | 1.47 (.53) | 1.32 (0.59) | 1.38 (.57)
Cardiopulmonary bypass time (hours) [Mean (Standard Deviation); unit: hours] — The block occurred at the end of surgery, so in no way should have affected intraoperative surgical characteristics. The characteristics of surgery are therefore a baseline measure, not an outcome measure.
  hours | 1.85 (.62) | 1.78 (.73) | 1.78 (.68)
Total surgical time (hours) [Mean (Standard Deviation); unit: hours] — The block occurred at the end of surgery, so in no way should have affected intraoperative surgical characteristics. The characteristics of surgery are therefore a baseline measure, not an outcome measure.
  hours | 4.88 (1.15) | 4.6 (1.3) | 4.73 (1.21)
Intraoperative oral morphine equivalents (mg) [Mean (Standard Deviation); unit: mg] — The block occurred at the end of surgery, so in no way should have affected intraoperative surgical characteristics. The characteristics of surgery are therefore a baseline measure, not an outcome measure.
  mg | 297.44 (65.13) | 276.64 (102.9) | 287.04 (86.05)

OUTCOME MEASURES:

1. Primary Outcome: Pain Scores at Rest Within the First 24 Hours After Extubation
Description: Measured by area under the curve (AUC) for pain scores gathered at 1, 3, 6, 12, 18, and 24 hours after extubation. To calculate the Area Under the Curve (AUC) for pain scores, pain intensity is plotted against time and the trapezoidal rule is used to approximate the area under the resulting curve. This AUC value represents the overall pain experience, considering both pain intensity and duration. Scale 0-240, with higher indicating a worse outcome. Units: Numeric rating score * hours.
Time Frame: 24 hours after extubation
Measure: Median (Inter-Quartile Range); unit: Numeric rating score * hours.
Arm/Group | Rectus Sheath Block With PIFB (Experimental Arm) | Rectus Sheath Block With PIFB (Placebo Arm)
Number analyzed (Participants) | 30 | 30
Numeric rating score * hours. | 79.25 [0 to 117] | 102 [65 to 120]

2. Primary Outcome: Pain Scores With Deep Breathing Within the First 24 Hours After Extubation
Description: as for outcome 1
Time Frame: 24 hours after extubation
Measure: Median (Inter-Quartile Range); unit: Numeric rating score * hours.
Arm/Group | Rectus Sheath Block With PIFB (Experimental Arm) | Rectus Sheath Block With PIFB (Placebo Arm)
Number analyzed (Participants) | 30 | 30
Numeric rating score * hours. | 141.5 [97 to 159.5] | 144 [90 to 160]

3. Primary Outcome: Total Cumulative Opioid Consumption
Description: Total cumulative opioid consumption at 24 hours
Time Frame: 24 hours post-operatively
Measure: Median (Inter-Quartile Range); unit: Oral morphine equivalents (mg)
Arm/Group | Rectus Sheath Block With PIFB (Experimental Arm) | Rectus Sheath Block With PIFB (Placebo Arm)
Number analyzed (Participants) | 30 | 30
Oral morphine equivalents (mg) | 55.25 [42.5 to 97.5] | 58.75 [42.5 to 91.5]

4. Primary Outcome: Total Cumulative Opioid Consumption
Description: Total cumulative opioid consumption at 48 hours
Time Frame: 48 hours post-operatively
Measure: Median (Inter-Quartile Range); unit: Oral morphine equivalents (mg)
Arm/Group | Rectus Sheath Block With PIFB (Experimental Arm) | Rectus Sheath Block With PIFB (Placebo Arm)
Number analyzed (Participants) | 30 | 30
Oral morphine equivalents (mg) | 96.75 [57.5 to 145] | 95 [55 to 130.25]

5. Secondary Outcome: Time From ICU Arrival to Liberation From Mechanical Ventilation
Description: Time from ICU arrival as measured by "anesthesia stop" to liberation from mechanical ventilation (extubation).
Time Frame: ICU arrival until extubation
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Rectus Sheath Block With PIFB (Experimental Arm) | Rectus Sheath Block With PIFB (Placebo Arm)
Number analyzed (Participants) | 30 | 30
hours | 3.87 [2.08 to 4.82] | 3.87 [2.63 to 4.80]

6. Secondary Outcome: Vital Capacity Change From Baseline on Incentive Spirometry
Description: Vital capacity change from baseline on incentive spirometry, measured as a percentage. An incentive spirometer was used to gather vital capacity (measured in mL).
Time Frame: 1 hour post-extubation
Population: 7 total patients did not have IS completed at 1 hour by ICU nursing due to either need for bipap/unknown reason.
Measure: Median (Inter-Quartile Range); unit: Percent of baseline IS
Arm/Group | Rectus Sheath Block With PIFB (Experimental Arm) | Rectus Sheath Block With PIFB (Placebo Arm)
Number analyzed (Participants) | 26 | 27
Percent of baseline IS | 0.25 [.17 to .29] | .24 [.18 to .34]

7. Secondary Outcome: Vital Capacity Change From Baseline on Incentive Spirometry
Description: as for outcome 6
Time Frame: 3 hours post-extubation
Measure: Median (Inter-Quartile Range); unit: Percent of baseline IS
Arm/Group | Rectus Sheath Block With PIFB (Experimental Arm) | Rectus Sheath Block With PIFB (Placebo Arm)
Number analyzed (Participants) | 30 | 30
Percent of baseline IS | .26 [.22 to .36] | .27 [.22 to .38]

8. Secondary Outcome: Vital Capacity Change From Baseline on Incentive Spirometry
Description: as for outcome 6
Time Frame: 12 hours post-extubation
Population: 3 total patients did not have IS completed at 12 hours by ICU nursing for unknown reasons
Measure: Median (Inter-Quartile Range); unit: Percent of baseline IS
Arm/Group | Rectus Sheath Block With PIFB (Experimental Arm) | Rectus Sheath Block With PIFB (Placebo Arm)
Number analyzed (Participants) | 28 | 29
Percent of baseline IS | .28 [.21 to .37] | .33 [.28 to .48]

9. Secondary Outcome: Vital Capacity Change From Baseline on Incentive Spirometry
Description: as for outcome 6
Time Frame: 24 hours post-extubation
Population: 7 total patients did not have IS completed at 24 hours by ICU nursing due to unknown reasons.
Measure: Median (Inter-Quartile Range); unit: Percent of baseline IS
Arm/Group | Rectus Sheath Block With PIFB (Experimental Arm) | Rectus Sheath Block With PIFB (Placebo Arm)
Number analyzed (Participants) | 26 | 27
Percent of baseline IS | .32 [.26 to .45] | .30 [.26 to .45]

10. Secondary Outcome: QoR-15 (Quality of Recovery) Score
Description: QoR-15 (Quality of Recovery) score is a 15 question survey asking patients about various aspects of their quality of recovery, including pain control, nausea, anxiety, depression, ability to eat, etc. The scale is 0-150, with higher scores indicating a better outcome.
Time Frame: 24 hours after extubation
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Rectus Sheath Block With PIFB (Experimental Arm) | Rectus Sheath Block With PIFB (Placebo Arm)
Number analyzed (Participants) | 30 | 30
score on a scale | 83 [70 to 106] | 79.5 [63 to 94]

11. Secondary Outcome: ICU Length of Stay
Description: ICU Length of Stay in hours, as measured by anesthesia stop until transfer out of the ICU.
Time Frame: Time from anesthesia stop to transfer out of ICU, typically 24 hours
Measure: Median (Inter-Quartile Range); unit: Hours
Arm/Group | Rectus Sheath Block With PIFB (Experimental Arm) | Rectus Sheath Block With PIFB (Placebo Arm)
Number analyzed (Participants) | 30 | 30
Hours | 20.69 [17.63 to 37.23] | 25.77 [22.28 to 45.22]

12. Secondary Outcome: Hospital Length of Stay
Description: Hospital Length of Stay in hours, as measured by anesthesia stop until discharge from the hospital.
Time Frame: Time from anesthesia stop to hospital discharge, typically one week
Measure: Median (Inter-Quartile Range); unit: Hours
Arm/Group | Rectus Sheath Block With PIFB (Experimental Arm) | Rectus Sheath Block With PIFB (Placebo Arm)
Number analyzed (Participants) | 30 | 30
Hours | 97.21 [89.16 to 135.89] | 97.31 [93.71 to 120.78]

ADVERSE EVENTS:
Time Frame: Each patient had adverse event data recorded through study completion and surgical follow-up, which was an average of one month.
Description: Each patient was seen POD 1 or 2 by the regional service to assess for complications. Also, study team members reviewed each patient's hospital course until the time of discharge to assess for complications, and OnCore was used to enroll patients in the study, which flagged the study team if the patient was seen/admitted (if documented in EPIC) post-discharge for any potential complications that could be reviewed. Each patient had adverse event data recorded through study completion.
Arm/Group | Rectus Sheath Block With PIFB (Experimental Arm) | Rectus Sheath Block With PIFB (Placebo Arm)
All-Cause Mortality (participants affected / at risk) | 0/30 | 1/32
Serious Adverse Events (participants affected / at risk) | 0/30 | 1/32
Other Adverse Events (participants affected / at risk) | 0/30 | 0/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rectus Sheath Block With PIFB (Experimental Arm) (N=30) | Rectus Sheath Block With PIFB (Placebo Arm) (N=32)
Acute right heart failure (Cardiac disorders) | 0 (0) | 1 (1) — A patient developed right heart failure postoperatively, requiring right ventricular assist device placement, which required removal from the study. The patient's clinical team and study independent monitor verified that this was not block-related.
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (32) — One patient expired within hours following surgery due to cardiac arrest that was determined to be the result of major surgical bleeding (cardiac). The patient's clinical team and study independent monitor verified that this was not block-related.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-09-30): https://cdn.clinicaltrials.gov/large-docs/49/NCT04908449/Prot_SAP_000.pdf
  • Informed Consent Form (2023-05-31): https://cdn.clinicaltrials.gov/large-docs/49/NCT04908449/ICF_001.pdf